CLINICAL TRIAL: NCT03860064
Title: Aneuploidy Rates of in Vitro Matured Oocytes
Acronym: IVM
Status: Completed | Type: Observational
Sponsor: IVI Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 1810-BCN-071-ME
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-07

CONDITIONS: Aneuploidy
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non intervention — Non

SUMMARY:
In general, nearly 85% of retrieved oocytes are mature and reproductively useful after the retrieval, whereas the remaining percentage are still at metaphase I or germinal vesicle stage (MI: 4% and GV: 11 %, respectively).

The objective of our study is to assess if immature oocytes co-cultured with autologous cumulus cells is a safer strategy than just leaving the oocytes in standard culture.

DETAILED DESCRIPTION:
Under controlled ovarian stimulation, patients with normal functional ovarian reserves produce a good number of oocytes at retrieval. However, in addition to quantity, oocyte maturity is an important variable for the success of reproductive technologies. In general, nearly 85% of retrieved oocytes are mature and reproductively useful, whereas the remaining percentage are still at metaphase I or germinal vesicle stage (MI: 4% and GV: 11 %, respectively). Due to the limited expectations held for in vitro maturation in said stimulated cycles, the rescue of immature oocytes is not widely used in current clinical practice and these oocytes are usually discarded due to the possibility of abnormal embryonic development or an increased rate of abortion.

The objective of our study is to assess if immature oocytes co-cultured with autologous cumulus cells is a safer strategy than just leaving the oocytes in standard culture.

ELIGIBILITY:
Inclusion Criteria:

* 18-35-year-old women
* BMI: >18 and < 30 kg/m2
* Normal female karyotype
* Normal uterus and ovaries at transvaginal ultrasound

Exclusion Criteria:

* > 35 years
* PCO syndrome carriers
* Null follicle aspiration
* History of chemotherapy or radiotherapy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Mature ooocytes from the same donors, will be used as control group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Aneuploidy rate | The moment that the PB is extruded (between 1 hour and 50 hours after the denudation)
  Aneuploidy rate of the PB

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Barcelona, Barcelona, Spain